CLINICAL TRIAL: NCT03562845
Title: Evaluation of the Clinical Consistency and Analytical Robustness of Immunobiogram® as an In Vitro Diagnostics Biotechnological Tool to Help Decision-making in Adjustment of Immunosuppressant Therapy for Renal Transplant
Brief Title: Evaluation of Immunobiogram® as a Tool in Adjustment of Immunosuppressant Therapy for Renal Transplant
Acronym: TRANSBIO
Status: Completed | Type: Observational
Sponsor: Biohope Scientific Solutions for Human Health, S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: BHP-IBG-2017-01
Record Dates: First submitted 2018-05-28; First posted 2018-06-20 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARM 1-Bad vs Good Clinical Evolution: This arm is intended to evaluate the correlation of Immunobiogram® sensitivity/resistance patterns with clinical prognosis as it may be judged at this moment considering clinical outcomes and immune-biomarker evolution in the past 12 to 18 months. Thus, it may confirm the BH-Pilot study findings. Renal transplant patients of two types will be included:
  * Patients who, over previous months, have had a bad clinical evolution, in which rejection mechanisms were involved
  * Patients with a good and stable clinical evolution
  IMBG sensitivity/resistance profiles will be compared amongst the two groups to evaluate the differences.
  Interventions: Other: NA-Observational only
- ARM 2-Stable Renal Transplant Patients: This arm is intended to evaluate robustness of Immunobiogram® as an IVD test. Thus, it will be performed intrasubject comparisons and inter-time evaluation of two sets of Immunobiogram® separated by 30+/- 10 days, each including three IMBG determinations (IMBGx3 - IMBGx3, the two sets separated by 30+/- 10 days). The intended evaluation will be to analyse the similarities between all IMBG tests performed, both between the same set and also between the two sets planned.
  Interventions: Other: NA-Observational only

INTERVENTIONS:
Other: NA-Observational only — NA-Observational only

SUMMARY:
The trial is an observational, multi-center study to determine if a new blood test (Immunobiogram®) done after renal transplant can help predict how well the immune system is working and responding to a new kidney. These blood tests could, in the future, potentially guide how doctors manage patient's anti-rejection medication.

DETAILED DESCRIPTION:
Rejection in renal transplants is a major problem unsolved in the long term, as 30-50% of patients lose their kidney due to rejection, or rejection mechanisms are involved elsewhere. One of the presumed key factors that may deliver such bad outcomes is the difficulties to personalise immunosuppressive treatment; a medical need that currently relies on immunosuppressive levels for some medications (pharmacokinetics), clinical guideline recommendations, adverse events profiles and some expensive biomarkers which are not widely used. Immunobiogram® (IMBG) is a tool that evaluates the sensitivity/resistance profile of patients to each of the most widely used and representative immunosuppressant drugs (IM). Thus, IMBG offers information that could become pivotal in clinical management of renal transplanted patients, if its potential benefits are proven. In this clinical study, a technology validation will be performed in which the robustness of the bioassay will be evaluated; and a correlation between the current clinical prognoses of each patient and resistance patterns will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Age > 25 years and < 70 years.
* Male and Female.
* Renal transplant performed at least 1 year before inclusion.

ARM 1:

* Bad clinical evolution: patients with renal dysfunction and positive biopsy to rejection OR significant increase in strength of DSA expressed as Luminex MFI. Specifically, the following two criteria must comply:

  * Renal function progressive deterioration, with significant creatinine increase of at least 15% for 18 months and/or proteinuria over > 500 mg/day or ratio protein/creatinine> 500 mg/g DE NOVO or increase in 50%.
  * Biopsy in the last 12 months that shows positive signs attributable to any kind of immunological response compatible with any type of rejection AND/OR at least 50% increase in strength of DSA expressed as Luminex MFI in comparison with previous determination and always at titers more than 3000UI.
* Good clinical evolution: patients without rejection episodes, negative DSA, stable renal function and no changes in treatment in the past 12 months. ALL the following criteria must apply

  * Stable renal function in the past 12 months
  * NO DSA titers
  * No history of previous rejection episodes
  * Stable immunosuppressive medication (No change in prednisone or MPA dose and tacrolimus dose with changes <20% of the dose) in the past 12 months

ARM 2:

* Stable renal function
* No DSA titers
* No history of previous rejection episodes
* Stable immunosuppressive medication (No change in prednisone or MPA dose and tacrolimus dose with changes <20% of the dose) at least in the past 18 months

Exclusion Criteria:

* Rejection of informed consent
* Active systemic infections that needed antimicrobial treatment in the past two months
* Active immune-based diseases with acute outbreaks in the past 12 months, despite immunosuppressive treatment
* Severe ischemia-reperfusion injury of current renal transplant with delayed graft function objectively evident at more than 20 days after transplant AND/OR kidney transplanted from a deceased, very elderly donor (>80 years)
* Double transplant (renal + another organ)
* HIV, HBV, HCV infection or other severe infectious diseases that prevent blood samples from being processed in a conventional laboratory
* Chronic Allograft Injury (CAI) unlikely related to immune processes, by the Investigator´s judgement
* Recurrent primary kidney disease

Ages: 25 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects <25 to < 70 years in age who have had a renal transplant performed at least one year before inclusion in the study
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the robustness of Immunobiogram® (IMBG) as an in vitro Diagnostic Bioassay to study the sensitivity/resistance patterns of Immunosuppressant drugs in Renal Transplantation | Baseline and 30 days
  Robustness of Immunobiogram® (IMBG) as an In Vitro Diagnostic Bioassay to study the sensitivity/resistance patterns of Immunosuppressant drugs in Renal Transplantation, evaluated as follows:
  * Immunobiogram® offers personal sensitivity/resistance patterns of Immunosuppressive Medications (IM), with a range of responses for each IM drug considering all patients included
  * Immunobiogram® shows intrasubject consistency in terms of similarity with a maximum +/- 20% of variation in the inhibitory dose/distance 50 (ID50), in the three IMBG performed on inclusion; and additionally, similar consistency must be observed in the last three IMBG performed one month after inclusion

SECONDARY OUTCOMES:
Evaluate intrasubject and inter-time consistency of Immunobiogram® | Baseline and 30 days
  Immunobiogram® shows intrasubject and inter-time consistency in terms of similarity with a maximum +/- 30% variation ID50, in the average response of the three IMBG performed on inclusion and the average response of the three IMBG performed one month after inclusion, provided that no significant clinical or immunological events happened during follow-up, as assessed with a specifically provided questionnaire and the Investigator´s judgement
Evaluate the correlation of Immunobiogram® sensitivity/resistance patterns with clinical evolution | Baseline
  ARM 1 describes the Immunobiogram® discrimination ranges based on the correlation with the results of sensitivity/resistance patterns to immunosuppressants as regards the trend of clinical progression in each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Pascual, MD, PhD, Principal Investigator — Parc du Salut Mar
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No